CLINICAL TRIAL: NCT00468702
Title: Postoperative Canadian Oral Anticoagulation Self-Management (Post-COAGS) Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD-0014; RD000000383-2007
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Cardiovascular Abnormalities
MeSH Terms: conditions — Cardiovascular Abnormalities

INTERVENTIONS:
Device: CoaguChek S

SUMMARY:
This study will measure the efficacy and safety of an early postoperative anticoagulation self-management program, using the CoaguChek S device, in patients undergoing mechanical valve replacements. Patients will be randomized into a study group (self-management) or a control group (physician management).

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-70 years of age;
* recipient of a mechanical heart valve (aortic and/or mitral), +/- CABG, +/- postoperative atrial fibrillation.

Exclusion Criteria:

* recipient of a bioprosthetic valve;
* post-operative thrombotic events;
* pre-operative utilization of oral anticoagulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Ottawa, Canada